CLINICAL TRIAL: NCT05872828
Title: Anxiety, Depression, Immune Function and Quality of Life Among Chinese Liver Cancer Patients in the COVID-19 Pandemic Era
Brief Title: Cross-sectional Study of Chinese Liver Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: The Nethersole School of Nursing (Other)
Responsible Party: Principal Investigator, Hua Yin, Principal Investigator, The Nethersole School of Nursing
Other Study IDs: SBRE-22-0307
Record Dates: First submitted 2023-03-23; First posted 2023-05-24 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Observational study. No intervention will be adopted.

SUMMARY:
The goal of this cross-sectional study is to investigate the prevalence and risk factors of anxiety and depression and their relationships with immune functions and quality of life among liver cancer patients in the COVID-19 pandemic era. The objectives of this study are:

1. To examine the prevalence of anxiety and depression among patients with liver cancer during the COVID-19 pandemic.
2. To identify risk factors associated with anxiety and depression among these patients.
3. To determine the association between anxiety, depression, immune function, and quality of life among liver cancer patients.

Participants will be asked to fill a digital questionnaire.

ELIGIBILITY:
Inclusion criteria

Participants must meet all the following criteria for study entry:

1. Aged 18 or older.
2. Participants have a confirmed diagnosis of liver cancer in the medical records.
3. Participants are able to communicate with Chinese. Exclusion criteria

Participants who meet any of the following criteria will be excluded from study entry:

1. Participant has multiple organ failure which makes him/her incapable to comply with the study protocol.
2. Participant has hepatic encephalopathy or severe mental disorder which makes him/her incapable of understanding the meanings of the questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients of liver cancer.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety score | Baseline
  Participants' anxiety status with HADS
Depression score | Baseline
  Participants' depression status with HADS

SECONDARY OUTCOMES:
Quality of life score (The EORTC QLQ-C30) | Baseline
  The European Organization for Research and Treatment of Cancer(EORTC) Quality of Life Questionnaire results. Scores range from 0 to 100. A higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Quality of life score (The EORTC QLQ-HCC18) | Baseline
  The Hepatocellular Carcinoma Module of The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire. Scores range from 0 to 100. A higher score represents a high level of symptomatology or problems.
Immune variables 1 | Baseline
  White blood cell counts (WBC). Collected from daily medical records.
Immune variables 2 | Baseline
  Total neutrophil count. Collected from daily medical records.
Immune variables 3 | Baseline
  Total lymphocyte count. Collected from daily medical records.
Immune variables 4 | Baseline
  Total monocyte count. Collected from daily medical records.
Immune variables 5 | Baseline
  Neutrophilic granulocyte percentage. Collected from daily medical records.
Immune variables 6 | Baseline
  Percentage of lymphocytes. Collected from daily medical records.
Immune variables 7 | Baseline
  Monocyte percentage. Collected from daily medical records.
Immune variables 8 | Baseline
  C-reactive protein (CRP). Collected from daily medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Yin, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Zhuhai People's Hospital, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Al-Quteimat OM, Amer AM. The Impact of the COVID-19 Pandemic on Cancer Patients. Am J Clin Oncol. 2020 Jun;43(6):452-455. doi: 10.1097/COC.0000000000000712. PMID 32304435
- [Background] Amiri S, Behnezhad S. Cancer Diagnosis and Suicide Mortality: A Systematic Review and Meta-Analysis. Arch Suicide Res. 2020;24(sup2):S94-S112. doi: 10.1080/13811118.2019.1596182. Epub 2019 May 9. PMID 30955459
- [Background] Antoni MH, Lechner S, Diaz A, Vargas S, Holley H, Phillips K, McGregor B, Carver CS, Blomberg B. Cognitive behavioral stress management effects on psychosocial and physiological adaptation in women undergoing treatment for breast cancer. Brain Behav Immun. 2009 Jul;23(5):580-91. doi: 10.1016/j.bbi.2008.09.005. Epub 2008 Sep 20. PMID 18835434
- [Background] Ayubi E, Bashirian S, Khazaei S. Depression and Anxiety Among Patients with Cancer During COVID-19 Pandemic: A Systematic Review and Meta-analysis. J Gastrointest Cancer. 2021 Jun;52(2):499-507. doi: 10.1007/s12029-021-00643-9. Epub 2021 May 5. PMID 33950368
- [Background] Blazeby JM, Currie E, Zee BC, Chie WC, Poon RT, Garden OJ; EORTC Quality of Life Group. Development of a questionnaire module to supplement the EORTC QLQ-C30 to assess quality of life in patients with hepatocellular carcinoma, the EORTC QLQ-HCC18. Eur J Cancer. 2004 Nov;40(16):2439-44. doi: 10.1016/j.ejca.2004.06.033. PMID 15519517
- [Background] Cao MD, Wang H, Shi JF, Bai FZ, Cao MM, Wang YT, Yan XX, Wang L, Huang Z, Ren JS, Zhao JJ, Dai M, Qu CF, Chen WQ. [Disease burden of liver cancer in China: an updated and integrated analysis on multi-data source evidence]. Zhonghua Liu Xing Bing Xue Za Zhi. 2020 Nov 10;41(11):1848-1858. doi: 10.3760/cma.j.cn112338-20200306-00271. Chinese. PMID 33297650
- [Background] Cao W, Li J, Hu C, Shen J, Liu X, Xu Y, Ye Z. Symptom clusters and symptom interference of HCC patients undergoing TACE: a cross-sectional study in China. Support Care Cancer. 2013 Feb;21(2):475-83. doi: 10.1007/s00520-012-1541-5. Epub 2012 Jul 20. PMID 23010958
- [Background] Chen G, Wu Q, Jiang H, Zhang H, Peng J, Hu J, Chen M, Zhong Y, Xie C. Fear of disease progression and psychological stress in cancer patients under the outbreak of COVID-19. Psychooncology. 2020 Sep;29(9):1395-1398. doi: 10.1002/pon.5451. Epub 2020 Jul 14. No abstract available. PMID 32596867
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Cheng C, Chan NY, Chio JH, Chan P, Chan AO, Hui WM. Being active or flexible? Role of control coping on quality of life among patients with gastrointestinal cancer. Psychooncology. 2012 Feb;21(2):211-8. doi: 10.1002/pon.1892. Epub 2010 Dec 19. PMID 22271542
- [Background] Cheng HH, Kamarck TW, Gianaros PJ, Roecklein KA, Vanegas Y, Tsung A, Geller DA, Marsh JW, Ahmed NS, Steel JL. Socioeconomic disparities of depressive symptoms and cytokines in hepatocellular carcinoma. Psychooncology. 2019 Aug;28(8):1624-1632. doi: 10.1002/pon.5127. Epub 2019 Jun 18. PMID 31119824
- [Background] Chu TL, Yu WP, Chen SC, Peng HL, Wu MJ. Comparison of differences and determinants between presence and absence of sleep disturbance in hepatocellular carcinoma patients. Cancer Nurs. 2011 Sep-Oct;34(5):354-60. doi: 10.1097/NCC.0b013e3182037bf3. PMID 21242769
- [Background] Chung MH, Wang SY, Lin CC. Symptom Clusters and Impact of Fatigue and Sleep Disturbance on Symptom Experiences of Hepatoma Patients in Taiwan. Cancer Nurs. 2017 Sep/Oct;40(5):403-411. doi: 10.1097/NCC.0000000000000417. PMID 27472191
- [Background] Dantzer R. Neuroimmune Interactions: From the Brain to the Immune System and Vice Versa. Physiol Rev. 2018 Jan 1;98(1):477-504. doi: 10.1152/physrev.00039.2016. PMID 29351513
- [Background] Dinarello CA. Proinflammatory cytokines. Chest. 2000 Aug;118(2):503-8. doi: 10.1378/chest.118.2.503. PMID 10936147
- See also: Quality of life questionnaires: EORTC QLQ-C30 & EORTC QLQ-HCC18. — http://qol.eortc.org/.